CLINICAL TRIAL: NCT02616679
Title: Cognitive Detection of Preclinical AD: Validation Using Biomarkers
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 13-00706
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Any remaining blood specimens will be retained indefinitely for future use by the Center for Cognitive Neurology (CCN) at NYU Langone Medical Center. Some samples may also be sent to Janssen Research & Development, LLC for potential future research use. Potential future research use by study investigators or collaborators will include possible discovery of novel biomarkers associated with increased AD risk, and study of validity of the use of such markers in preclinical AD. True genetic testing will not be done on these samples.
  Subjects may decline to have their samples stored for future use by checking the applicable box on the informed consent form. Subjects who agreed to have their samples stored for future use may revoke this permission.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitively Normal: Participants will be deemed cognitively normal based on criteria set forth by the National Alzheimer's Disease Coordinating Center/Alzheimer's Disease Centers (ADCC/ADC).
- Amnestic Mild Cognitive Impairment (aMCI): Participants will be deemed aMCI based on criteria set forth by the National Alzheimer's Disease Coordinating Center/Alzheimer's Disease Centers (ADCC/ADC).

SUMMARY:
The current study aims to validate several novel cognitive tasks expected to be sensitive to brain impairment in specific anatomic regions affected in preclinical Alzheimer's disease(pAD). The tasks are validated in 60 cognitively and clinically normal participants ages 60 - 85, inclusive, against reasonably well-established biomarkers of Alzheimer's disease, including 1) simultaneous positron emission tomography (PET) [18F]Flutemetamol amyloid and CT imaging and 2) to the extent data is available from other studies, participants' brain MRI and cerebral spinal fluid (CSF) amyloid and tau.

DETAILED DESCRIPTION:
Biomarkers, such as amyloid deposition, and Hipp volume loss, and low Aβ and high pTau in CSF, are useful for identifying cognitively normal (CN) elderly who are likely have early AD pathology ("preclinical AD"). However, they are invasive and/or expensive. The goal of the current study is to develop and validate cognitive proxies of AD biomarkers by using cognitive tasks that are dependent on brain regions impaired by very early AD pathology. If successful, these tasks will provide a non-invasive and cost-effective way to identify and track change in CN individuals at high risk for progressing to mild cognitive impairment (MCI) and dementia stages of AD and thus will facilitate future prevention trials in pAD.

Subjects will attend three study visits. During the first study visit, subjects will have eligibility criteria confirmed, have a blood sample drawn, and complete about half of the cognitive tasks. The second visit, which will occur within one week of visit one, will involve completion of the remaining cognitive tasks. Subjects will also be asked to have a PET-CT scan during visit three (to occur within 3 months of visits 1 and 2).

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment as a participant in the NYU Alzheimer's Disease Center (ADC) and completion of the ADC Clinical Evaluation within the past year.
* Clinical diagnosis of "cognitively normal" or "amnestic mild cognitive impairment" based on recent (within 1 year) consensus meeting cross-referenced with standard neuropsychological scores.
* Normal or corrected-to-normal vision and hearing (able to see images on computer screen and hear auditory events delivered through the computer speaker).

Exclusion Criteria:

* Significant history of mental illness, drug or alcohol abuse; severe trauma preventing normal use of dominant hand (needed to move the mouse cursor); clinical depression (unless medically controlled); other neurologic conditions (i.e. stroke), or learning disability; ophthalmologic/visual problems that prevent viewing a computer screen at a normal distance (such as legal blindness, detached retinas, occlusive cataracts).
* Lack of capacity to give informed consent and no legally authorized representative to provide consent.
* Having pacemakers, aneurysm clips, cochlear implants, or metal/foreign objects in body and therefore, unable to receive MRI.
* Pregnancy, breastfeeding or planning to have a baby.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants will be elderly individuals who are participating in ongoing clinical research at the NYU CCN, including at the ADC and the Center for Brain Health (CBH). Participants may also be recruited through community outreach or referrals from other centers. Cognitively normal (CN) participants and participants with amnestic mild cognitive impairment (aMCI) will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2020-08-12 (Actual)

PRIMARY OUTCOMES:
Correlation of composite score on cognitive tests with biomarkers | 3 months
  The overall score on the cognitive tests will be correlated via a linear regression with biomarker data collected during the study. Each biomarker will be regressed individually. Biomarker data includes: MRI hippocampus (hipp) volume, entorhinal cortex (EC) volume, EC standard uptake value ratios (SUVRs), Hipp SUVR, precuneus (PCu) SUVR, PET-[18F] Flutemetamol SUVR, CSF Aβ and tau levels, levels of diffusion tensor imaging mean diffusivity, and levels of fractional anisotropy.

SECONDARY OUTCOMES:
Presence of ApoE allele | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sadowski, PhD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU Langone Medical Center, New York, New York, United States